CLINICAL TRIAL: NCT02931435
Title: Radiofrequency For The Treatment Of Chronic Knee Pain Following Total Knee Arthroplasty: A Double-Blind Randomized Controlled Pilot Study
Brief Title: Radiofrequency For Chronic Knee Pain Post-Arthroplasty
Acronym: DEFIANT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Randall Brewer, MD, CPI (Other)
Collaborators: Abbott Medical Devices (Industry); Abbott (Industry)
Responsible Party: Sponsor-Investigator, Randall Brewer, MD, CPI, Medical Director, Principal Investigator, Willis-Knighton River Cities Clinical Research Center
Organization: Willis-Knighton River Cities Clinical Research Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GENRF
Record Dates: First submitted 2016-10-05; First posted 2016-10-13 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Chronic Knee Pain; Osteoarthritis, Knee
Keywords: Genicular Radiofrequency Ablation; Knee Arthroplasty, Total
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Nerve Block; Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nerve Block with Radiofrequency Ablation (Active Comparator): A 10 cm 18-gauge RF cannula with a 10 mm active tip will be placed at the superior lateral, superior medial, and inferior medial nerve positions under fluoroscopic guidance. Sensory stimulation at 50 Hz will be performed to identify nerve position and to assure no motor nerves will be ablated. Lidocaine (2 ml of 2%) will be administered in each location prior to RF generator activation.
  Interventions: Procedure: Nerve Block with Radiofrequency Ablation
- Nerve Block with Sham Radiofrequency Ablation (Sham Comparator): A 10 cm 18-gauge RF cannula with a 10 mm active tip will be placed at the superior lateral, superior medial, and inferior medial nerve positions under fluoroscopic guidance.Control patients will undergo the same procedure without RF generator activation. Sensory stimulation at 50 Hz will be performed to identify nerve position and to assure no motor nerves will be ablated. Lidocaine (2 ml of 2%) will be administered in each location prior to RF generator sham activation.
  Interventions: Procedure: Nerve Block with Sham Radiofrequency Ablation

INTERVENTIONS:
Procedure: Nerve Block with Radiofrequency Ablation — Ablation of the genicular nerves of the knee by radiofrequency
  Arms: Nerve Block with Radiofrequency Ablation
Procedure: Nerve Block with Sham Radiofrequency Ablation — Genicular radiofrequency of the knee without neurotomy
  Arms: Nerve Block with Sham Radiofrequency Ablation

SUMMARY:
Chronic knee osteoarthritis (OA) is one of the most common diseases with increasing prevalence in advanced age. Knee OA results in movement restriction, sleep disturbance, and disability. Total knee arthroplasty (TKA) is employed often in the symptomatic treatment of knee OA. It has been estimated that 3.4 million TKAs will be performed in the year 2030 in the United States alone. Many studies report rewarding outcomes for patients, but other research shows there are many patients that remain dissatisfied post-arthroplasty.

The purpose of this study is to evaluate whether genicular radiofrequency ablation can relieve chronic post-arthroplasty knee pain.

DETAILED DESCRIPTION:
Chronic knee osteoarthritis (OA) is one of the most common diseases with increasing prevalence in advanced age. Knee OA results in movement restriction, sleep disturbance, and disability. Total knee arthroplasty (TKA) is employed often in the symptomatic treatment of knee OA. It has been estimated that 3.4 million TKAs will be performed in the year 2030 in the United States alone. Many studies report rewarding outcomes for patients, but other research shows there are many patients that remain dissatisfied post-arthroplasty.

As the prevalence of knee arthroplasty increases, so does the frequency of revisions. It has been found that 20% of patients reporting painful knee arthroplasties were not able to be diagnosed with a specific cause and were therefore referred to a pain specialist. Pharmacologic therapy and non-surgical interventions are often employed with minimal benefit to the patient's level of disability as indicated by clinical evidence.

Genicular radiofrequency ablation seems to be a safe, effective and minimally invasive therapy for chronic knee OA patients who have had a positive diagnostic block. No study has determined whether genicular radiofrequency ablation can relieve chronic post-arthroplasty knee pain. The investigators propose to examine the effect of genicular radiofrequency ablation in chronic post-arthroplasty knee pain in patients who respond positively to diagnostic nerve blocks.

ELIGIBILITY:
Inclusion Criteria:

* Study candidate must provide written informed consent.
* Must be ≥ 50 years of age at the time of consent
* Chronic knee pain despite total knee arthroplasty at least 6 months prior to consent
* Orthopedic evaluation indicating no further surgery is warranted
* Stable pain medication regimen for 30 days prior to baseline visit
* Knee pain is primary pain complaint

Exclusion Criteria:

* Acute knee pain
* Connective tissue disorders affecting the knee
* Serious neurologic or psychiatric disorders that would affect the outcome of the study as determined by the Principal Investigator
* Steroid or hyaluronic acid injections into the affected knee in the past 3 months
* Confounding pain conditions of the index leg that may affect medication requirements or study outcomes

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-12; Primary Completion 2018-11-20 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Mean difference in knee pain intensities as indicated on the Visual Analog Scale | Baseline and 6 weeks post-radiofrequency ablation

SECONDARY OUTCOMES:
Change in Visual Analog Score of average knee pain | Baseline to 1 week, 6 weeks, and 12 weeks
Change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Baseline to 1 week, 6 weeks, and 12 weeks
Change in Knee Injury and Osteoarthritis Outcome Score (KOOS) | Baseline to 1 week, 6 weeks, and 12 weeks
Change of Patient Global Assessment | Baseline to 1 week, 6 weeks, and 12 weeks
Satisfaction with Radiofrequency Procedure | Baseline to 1 week, 6 weeks, and 12 weeks
Rate of procedure-related Adverse Events | From informed consent through study completion, up to 20 weeks
Rate of Serious Adverse Events | From informed consent through study completion, up to 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Randall Brewer, MD, Principal Investigator — WK River Cities Clinical Research Center
Locations (1):
- WK River Cities Clinical Research Center, Shreveport, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Background] Nikolaou VS, Chytas D, Babis GC. Common controversies in total knee replacement surgery: Current evidence. World J Orthop. 2014 Sep 18;5(4):460-8. doi: 10.5312/wjo.v5.i4.460. eCollection 2014 Sep 18. PMID 25232522
- [Background] Choi WJ, Hwang SJ, Song JG, Leem JG, Kang YU, Park PH, Shin JW. Radiofrequency treatment relieves chronic knee osteoarthritis pain: a double-blind randomized controlled trial. Pain. 2011 Mar;152(3):481-487. doi: 10.1016/j.pain.2010.09.029. Epub 2010 Nov 4. PMID 21055873
- [Background] Al-Hadithy N, Rozati H, Sewell MD, Dodds AL, Brooks P, Chatoo M. Causes of a painful total knee arthroplasty. Are patients still receiving total knee arthroplasty for extrinsic pathologies? Int Orthop. 2012 Jun;36(6):1185-9. doi: 10.1007/s00264-011-1473-6. Epub 2012 Jan 11. PMID 22234706